CLINICAL TRIAL: NCT04372147
Title: Embolization of the Middle Meningeal Artery for the Prevention of Chronic Subdural Hematoma Recurrence in High Risk Patients, a Randomized Controlled Trial
Brief Title: Embolization of the Middle Meningeal Artery for the Prevention of Chronic Subdural Hematoma Recurrence in High Risk Patients (EMPROTECT)
Acronym: EMPROTECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP180574
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-01

CONDITIONS: Chronic Subdural Hematoma; At Risk of Post-operative Recurrence; Burr-hole Surgery
Keywords: Chronic Subdural Hematoma; Burr-Hole Surgery; Recurrence; Middle Meningeal Artery; Embolization
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Recurrence

STUDY DESIGN:
Intervention Model Description: multicenter open label randomized controlled trial. Eligible patients will be assigned either to the intervention or a control arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): MMA embolization procedure within 7 days of the burr-hole surgery in addition to standard medical care
  Interventions: Procedure: MMA embolization
- control group (No Intervention): standard medical care

INTERVENTIONS:
Procedure: MMA embolization — Patients in the intervention group will undergo a CT angiography scan of the supra aortic trunks, followed by MMA embolization procedure within 7 days of the burr-hole surgery in addition to standard medical care
  Arms: intervention group

SUMMARY:
Standard of care for the management of symptomatic chronic subdural hematomas (SDHs) is neurosurgical burr-hole evacuation followed by drainage. Post-operative recurrence rates may be as high as 10 to 20 %. In particular, recurrence rate increases with antiplatelet and anticoagulant therapy. Middle meningeal artery (MMA) embolization has been proposed as a novel treatment of chronic SDH. The aim of this study is to assess the efficacy of MMA embolization in reducing the risk of chronic SDH recurrence at 6 months after burr-hole surgery as compared with standard medical post-operative treatment in patients at high risk of post-operative recurrence.

DETAILED DESCRIPTION:
Introduction: chronic SDHs are some of the most frequently encountered neurosurgical emergencies. The gold standard treatment of symptomatic chronic SDHs is burr-hole surgery followed by temporary closed system drainage. Post-operative recurrence rates may be as high as 10 to 20% and are a major source of morbidity and repeated surgery. MMA embolization is a promising minimally invasive procedure recently proposed as a treatment of chronic SDH. It is hypothesized that post-operative MMA embolization may reduce recurrence rate in patients at high risk of recurrence.

Aims: the primary objective of the trial is to assess the efficacy of MMA embolization in reducing the risk of chronic SDH recurrence at 6 months after burr-hole surgery as compared with standard medical treatment in patients at high risk of post-operative recurrence. Secondary objectives include evaluating the impact of post-operative MMA embolization on rate of recurrence requiring new surgery (at 6 months), rate of functional dependency (at 1 and 6 months) , mortality (at 1 and 6 months) , cumulative hospital stay duration, related to the SDH, and complication rate at 6 months.

Methods: multicenter open label randomized controlled trial. Eligible patients will be assigned either to the intervention or a control arm through blocked randomization with randomblock sizes and stratified on the center, antiplatelet/anticoagulant therapy and unilateral vs bilateral SDH. Patients in the intervention group will undergo a CT angiography scan of the supra aortic trunks, followed by MMA embolization procedure within 7 days of the burr-hole surgery in addition to standard medical care. Patients in the control group will receive standard medical care only. Outcomes will be evaluated at 1 and 6 months. The primary outcome measure will be the rate of chronic SDH recurrence 6 months after index burr-hole surgery, as defined bellow. In order to demonstrate a decrease in recurrence rate from 15 to 5% between the intervention and control arms with a power of 80%, bilateral global alpha risk of 5%, with two planned sequential tests according to the method of Lan & Demets, and 20% patients lost to follow-up, 342 patients are required, 171 in each arm. The primary outcome will be analyzed according to intention to treat.

ELIGIBILITY:
Inclusion Criteria:

Patient:

* Aged ≥ 18 years
* Operated for a SDH recurrence or operated for a first episode of SDH if at least one of the following recurrence risk factors is present:
* Chronic alcoholism defined by a daily alcohol consumption > 30g/day
* Or liver cirrhosis
* Or antiplatelet therapy
* Or anticoagulant therapy
* Or thrombocytopenia with a platelet count < 100 x10(3) per µL
* Or surgery without use of external drain
* With affiliation to a social security scheme
* Having signed an informed consent form or for whom a delegate close relative or a support person has signed an informed consent

Exclusion Criteria:

* SDH evacuation by craniotomy or twist-drill craniostomy rather than burr-hole surgery
* Beyond 7 days after the index surgery (surgery for recurrent SDH or first surgery in case of a risk factor as indicated in the inclusion criteria)
* Functionally dependant patient with an mRS score ≥ 4 before the SDH
* Patient with a life expectancy < 6 months
* Patient with renal failure as defined by a creatinine clearance < 30 ml/min
* Pregnancy
* History of allergy to a iodinated contrast agent
* Procedure deemed unachievable under local anesthesia (because of patient agitation or discomfort for instance) in a patient with a contraindication to both conscious sedation and general anesthesia.
* Patient refusal
* Patient for whom follow-up is deemed problematic (living abroad or homeless for instance )
* Patients under legal guardianship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
SDH recurrence | 6 months
  Rate of chronic subdural hematoma (SDH) recurrence 6 months after index burr-hole surgery, defined as:
  * Reappearance of a homolateral SDH with a midline shift > 5mm or a symptomatic homolateral SDH, including leading to death
  * Or, the presence of a homolateral SDH > 10mm in maximal thickness on the 6 months control head CT scan
  * Or, the need for repeated surgery for a homolateral SDH recurrence
  * Or, the need for a new hospital admission in relation to a homolateral SDH recurrence

SECONDARY OUTCOMES:
repeated surgery | 6 months
  - Rate of repeated surgery for a homolateral SDH recurrence during the 6 months follow-up period
disability and dependency | 1 and 6 months
  - Rate of disability and dependency at 1 and 6 months, defined by a modified Rankin Scale (mRS) score ≥ 4.
  The mRS is an ordered scale coded from 0 (no symptoms at all) through 5 (severe disability) 6 (death)
mortality | 1 and 6 months
  - Mortality rate at 1 and 6 months
hospital stay | 6 months
  - Total cumulative duration of hospital stay, during the 6 months follow-up period, directly or indirectly related to the SDH
complication rates | 6 months
  - Minor and major embolization procedure-related complication rates

CONTACTS AND LOCATIONS:
Overall Officials: Eimad Shotar, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (12):
- France (12):
  - Hôpital d'instruction des armées de Percy, Clamart
  - Hôpital Beaujon, Clichy
  - Hôpital Henri-Mondor, Créteil
  - CHU Lille (Hôpital Roger Salengro), Lille
  - CHU de Limoges, Limoges
  - Hôpital Nord (CHU MARSEILLE), Marseille
  - CHU de Marseille, Marseille
  - Hôpital Lariboisière, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Sainte Anne, Paris
  - Fondation Rothschild, Paris
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Shotar E, Mathon B, Salle H, Rouchaud A, Mounayer C, Bricout N, Lejeune JP, Janot K, Amelot A, Naggara O, Roux A, Goutagny S, Guedon A, Houdart E, Brunel H, Hak JF, Troude L, Dufour H, Bernat AL, Tuilier T, Bresson D, Apra C, Fouet M, Escalard S, Chauvet D, Premat K, Lebbah S, Dechartres A, Clarencon F; EMPROTECT Investigators. Meningeal Embolization for Preventing Chronic Subdural Hematoma Recurrence After Surgery: The EMPROTECT Randomized Clinical Trial. JAMA. 2025 Jul 8;334(2):127-135. doi: 10.1001/jama.2025.7583. PMID 40471557
- [Derived] Shotar E, Mathon B, Rouchaud A, Mounayer C, Salle H, Bricout N, Lejeune JP, Janot K, Zemmoura I, Naggara O, Roux A, Goutagny S, Guedon A, Brunel H, Troude L, Dufour H, Bernat AL, Tuilier T, Bresson D, Apra C, Fouet M, Escalard S, Chauvet D, Baptiste A, Lebbah S, Dechartres A, Clarencon F; EMPROTECT collaboration. Embolization of the middle meningeal artery for the prevention of chronic subdural hematoma recurrence in high-risk patients: a randomized controlled trial-the EMPROTECT study protocol. J Neurointerv Surg. 2024 Dec 26;17(e1):e172-e177. doi: 10.1136/jnis-2023-021249. PMID 38307722